CLINICAL TRIAL: NCT06117722
Title: ESTIA: TorasEmide Induced Effect on Quality of Life and Clinical parameterS in paTients With chronIc heArt Failure Receiving Eplerenone. Multicenter, Non-interventional, Prospective, Observational Clinical Study.
Brief Title: TorasEmide Induced Effect on QoL and Clinical parameterS in paTients With chronIc heArt Failure Receiving Eplerenone.
Acronym: ESTIA
Status: Recruiting | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-TOREPL-EL-184
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Eplerenone torasemide in chronic heart failure — Heart Failure patients treated with eplerenone and torasemide

SUMMARY:
Heart failure (HF) is a multisystemic disorder characterized by marked disturbances in the physiology of the circulatory system and a multitude of structural and functional changes in the myocardium that adversely affect the systolic function and diastolic filling of the heart. Heart failure is not a single pathologic diagnosis, but a clinical syndrome consisting of cardiac symptoms (eg, dyspnea, edema of the lower extremities, and fatigue) that may be accompanied by signs (eg, increased jugular venous pressure and peripheral edema).The diagnosis of CKD becomes more likely in patients with a history of myocardial infarction (MI), arterial hypertension, coronary artery disease (CHD), diabetes mellitus, alcohol abuse, chronic kidney disease (CKD), cardiotoxic chemotherapy, and in patients with a family history of cardiomyopathy or of sudden death. The diagnosis of HF requires the presence of HF symptoms and/or signs and objective evidence of cardiac dysfunction.

The main symptoms of HF are symptoms such as shortness of breath at rest or during exercise, difficulty breathing (dyspnea), rapid breathing (tachypnea), difficulty breathing when bending over (bendopnea), orthopnea, paroxysmal nocturnal dyspnea, fatigue , weight gain or weight loss, swelling (of the extremities, scrotum or elsewhere), wheezing, palpitations, syncope, history of Cheyne Stokes breathing during sleep (often reported by the family rather than the patient), cough, drowsiness.

The simplest terminology used to describe HF severity is the New York Heart Association (NYHA) functional classification based on symptom severity and physical activity.

In Greece, it is estimated that the number of patients suffering from HF is 200,000.

In the vast majority of cases, transthoracic echocardiography is the initial cardiac imaging test used to evaluate patients with newly diagnosed or suspected heart failure. Echocardiography is particularly suitable for the evaluation of myocardial structure and function, valvular function and hemodynamic parameters .

DETAILED DESCRIPTION:
Eplerenone is more specific in blocking aldosterone and therefore causes less gynecomastia. Eplerenone is indicated in addition to standard therapy including β-blockers to reduce the risk of cardiovascular mortality and morbidity in stable patients with left ventricular dysfunction (LVEF ≤40%) and clinical evidence of heart failure after recent myocardial infarction. In addition, eplerenone is indicated in standard optimal therapy to reduce the risk of cardiovascular mortality and morbidity in adult patients with NYHA class II (chronic) HF and with left ventricular systolic dysfunction (LVEF ≤ 30%).

Caution should be exercised when MRAs are used in patients with renal impairment and those with serum potassium concentrations >5.0 mmol/L.

Diuretics are drugs that are recommended or should be considered in selected HF patients with reduced ejection fraction. The goal of diuretic therapy is to achieve and maintain euvolemia with the lowest dose of diuretics.

Loop diuretics are recommended to reduce signs and/or symptoms of congestion in patients with HFrEF.

Transition to oral therapy should begin when the patient's clinical condition is stable .

Torasemide, one of the loop diuretics, is indicated in the treatment of edema due to congestive heart failure. The usual starting dose is 10 or 20 mg once a day. If the diuretic response is inadequate, the dose should be approximately doubled until an adequate response is achieved .

Among the potential advantages of torasemide in the treatment of HF are its beneficial pharmacological properties, which make it more suitable for the management of congestion ).

Torasemide may be less susceptible to diuretic resistance, has a prolonged half-life (3.5 hours), prolonged duration of effect (6-16 hours), and is less prone to hypokalemia .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with a diagnosis of Chronic Heart Failure (CHF)
* Patients who are on treatment with torasemide added on to eplerenone treatment, from 1 to 7 days before study initiation.
* Patients who are able to provide informed consent and follow study procedures and requirements.

Exclusion Criteria:

* Patients with hypersensitivity to the active substance of torasemide, sulfonylureas or to any of the excipients mentioned in torasemide SmPC.
* Patients with renal failure with anuria.
* Patients in hepatic coma, or pro-coma.
* Patients with intolerance to galactose, complete lactase deficiency or glucose-galactose malabsorption.
* Patients with hypotension.
* Patients with cardiac arrhythmias.
* Patients with parallel treatment with aminoglycosides or cephalosporins.
* Patients with kidney dysfunction due to drugs that cause kidney damage.
* The addition during the study of other drugs with a direct effect on diuresis (such as other diuretics or SGLT2 inhibitors).
* Patients who are unable to comply with the study protocol procedures and requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of Chronic Heart Failure (CHF) who are on treatment with torasemide added on to eplerenone treatment, from 1 to 7 days before study initiation.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure (MLHF) | 6 months
  The change in the disease specific questionnaire - Minnesota Living with Heart Failure (MLHF) - score from baseline to 6 months of treatment and between the visits.

SECONDARY OUTCOMES:
CHQ-SAS (Chronic Heart failure Questionnaire - Self Administered format, Standardized questions) | 6 months
  Changes from baseline in the CHQ-SAS (Chronic Heart failure Questionnaire - Self Administered format, Standardized questions) to assess the degree of dyspnoea, between the visits and at 6 months from treatment initiation.
  Changes from baseline in patients' New York Heart Association (NYHA) classification between the visits and at 6 months.
New York Heart Association (NYHA) classification | 6 months
  Changes from baseline in patients' New York Heart Association (NYHA) classification between the visits and at 6 months.
Morisky Medication Adherence Scale (MMAS-8) | 6 months
  The score of the 8-item Morisky Medication Adherence Scale (MMAS-8) at 3 and 6 months from treatment initiation and its change between visits.
Body weight | 6 months
  The change in patients' body weight from baseline, between the visits and at 6-months from treatment initiation.
Dosage scheme | 6 months
  The record of torasemide titration.
Number of Adverse Events | 6 months
  The record of Adverse Events during the study conduct.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Ginis, MD, Study Director — Elpen Pharmaceutical Industry
Locations (1):
- ATTIKON University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diwan, A. &. (2019). SECTION I Basic Mechanisms of Heart Failure. Heart Failure: A Companion to Braunwald's Heart Disease, 1.
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Lam CSP, Voors AA, Piotr P, McMurray JJV, Solomon SD. Time to rename the middle child of heart failure: heart failure with mildly reduced ejection fraction. Eur Heart J. 2020 Jul 1;41(25):2353-2355. doi: 10.1093/eurheartj/ehaa158. No abstract available. PMID 32227233
- [Background] Mant J, Doust J, Roalfe A, Barton P, Cowie MR, Glasziou P, Mant D, McManus RJ, Holder R, Deeks J, Fletcher K, Qume M, Sohanpal S, Sanders S, Hobbs FD. Systematic review and individual patient data meta-analysis of diagnosis of heart failure, with modelling of implications of different diagnostic strategies in primary care. Health Technol Assess. 2009 Jul;13(32):1-207, iii. doi: 10.3310/hta13320. PMID 19586584
- [Background] Davie AP, Francis CM, Caruana L, Sutherland GR, McMurray JJ. Assessing diagnosis in heart failure: which features are any use? QJM. 1997 May;90(5):335-9. doi: 10.1093/qjmed/90.5.335. PMID 9205668
- [Background] Oudejans I, Mosterd A, Bloemen JA, Valk MJ, van Velzen E, Wielders JP, Zuithoff NP, Rutten FH, Hoes AW. Clinical evaluation of geriatric outpatients with suspected heart failure: value of symptoms, signs, and additional tests. Eur J Heart Fail. 2011 May;13(5):518-27. doi: 10.1093/eurjhf/hfr021. Epub 2011 Mar 19. PMID 21422000
- [Background] Kelder JC, Cramer MJ, van Wijngaarden J, van Tooren R, Mosterd A, Moons KG, Lammers JW, Cowie MR, Grobbee DE, Hoes AW. The diagnostic value of physical examination and additional testing in primary care patients with suspected heart failure. Circulation. 2011 Dec 20;124(25):2865-73. doi: 10.1161/CIRCULATIONAHA.111.019216. Epub 2011 Nov 21. PMID 22104551
- [Background] Caraballo C, Desai NR, Mulder H, Alhanti B, Wilson FP, Fiuzat M, Felker GM, Pina IL, O'Connor CM, Lindenfeld J, Januzzi JL, Cohen LS, Ahmad T. Clinical Implications of the New York Heart Association Classification. J Am Heart Assoc. 2019 Dec 3;8(23):e014240. doi: 10.1161/JAHA.119.014240. Epub 2019 Nov 27. PMID 31771438
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292
- [Background] Dunlay SM, Roger VL. Understanding the epidemic of heart failure: past, present, and future. Curr Heart Fail Rep. 2014 Dec;11(4):404-15. doi: 10.1007/s11897-014-0220-x. PMID 25182014
- [Background] Roth GA, Forouzanfar MH, Moran AE, Barber R, Nguyen G, Feigin VL, Naghavi M, Mensah GA, Murray CJ. Demographic and epidemiologic drivers of global cardiovascular mortality. N Engl J Med. 2015 Apr 2;372(14):1333-41. doi: 10.1056/NEJMoa1406656. PMID 25830423
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Meyer S, Brouwers FP, Voors AA, Hillege HL, de Boer RA, Gansevoort RT, van der Harst P, Rienstra M, van Gelder IC, van Veldhuisen DJ, van Gilst WH, van der Meer P. Sex differences in new-onset heart failure. Clin Res Cardiol. 2015 Apr;104(4):342-50. doi: 10.1007/s00392-014-0788-x. Epub 2014 Nov 15. PMID 25398254
- [Background] Brouwers FP, de Boer RA, van der Harst P, Voors AA, Gansevoort RT, Bakker SJ, Hillege HL, van Veldhuisen DJ, van Gilst WH. Incidence and epidemiology of new onset heart failure with preserved vs. reduced ejection fraction in a community-based cohort: 11-year follow-up of PREVEND. Eur Heart J. 2013 May;34(19):1424-31. doi: 10.1093/eurheartj/eht066. Epub 2013 Mar 6. PMID 23470495
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Cosin J, Diez J; TORIC investigators. Torasemide in chronic heart failure: results of the TORIC study. Eur J Heart Fail. 2002 Aug;4(4):507-13. doi: 10.1016/s1388-9842(02)00122-8. PMID 12167392
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Moradi M, Daneshi F, Behzadmehr R, Rafiemanesh H, Bouya S, Raeisi M. Quality of life of chronic heart failure patients: a systematic review and meta-analysis. Heart Fail Rev. 2020 Nov;25(6):993-1006. doi: 10.1007/s10741-019-09890-2. PMID 31745839
- [Background] Plakas S, Mastrogiannis D, Mantzorou M, Adamakidou T, Fouka G, Bouziou A, et al. Validation of the 8-Item Morisky Medication adherence scale in chronically Ill ambulatory patients in Rural Greece. Open J Nurs. 2016;06:158-69.
- [Background] Tan X, Patel I, Chang J. Review of the four item Morisky medication adherence scale (MMAS-4) and eight item Morisky Medication Adherence Scale (MMAS-8). Innov Pharm. 2014;5:11478.
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Krousel-Wood M, Islam T, Webber LS, Re RN, Morisky DE, Muntner P. New medication adherence scale versus pharmacy fill rates in seniors with hypertension. Am J Manag Care. 2009 Jan;15(1):59-66. PMID 19146365
- [Background] Morisky DE, DiMatteo MR. Improving the measurement of self-reported medication nonadherence: response to authors. J Clin Epidemiol. 2011 Mar;64(3):255-7; discussion 258-63. doi: 10.1016/j.jclinepi.2010.09.002. Epub 2010 Dec 8. No abstract available. PMID 21144706
- [Background] Martinez-Perez P, Orozco-Beltran D, Pomares-Gomez F, Hernandez-Rizo JL, Borras-Gallen A, Gil-Guillen VF, Quesada JA, Lopez-Pineda A, Carratala-Munuera C. Validation and psychometric properties of the 8-item Morisky Medication Adherence Scale (MMAS-8) in type 2 diabetes patients in Spain. Aten Primaria. 2021 Feb;53(2):101942. doi: 10.1016/j.aprim.2020.09.007. Epub 2021 Jan 25. PMID 33508739
- [Background] Gupta S, Goren A. Application of item response theory in validating the Morisky medication adherence scale in patients with hypertension. Value Health. 2013;16:A4.
- [Background] Naveiro-Rilo JC, Diez-Juarez DM, Romero Blanco A, Rebollo-Gutierrez F, Rodriguez-Martinez A, Rodriguez-Garcia MA. Validation of the Minnesota living with heart failure questionnaire in primary care. Rev Esp Cardiol. 2010 Dec;63(12):1419-27. doi: 10.1016/s1885-5857(10)70276-0. English, Spanish. PMID 21144402
- [Background] Behlouli H, Feldman DE, Ducharme A, Frenette M, Giannetti N, Grondin F, Michel C, Sheppard R, Pilote L. Identifying relative cut-off scores with neural networks for interpretation of the Minnesota Living with Heart Failure questionnaire. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6242-6. doi: 10.1109/IEMBS.2009.5334659. PMID 19965089
- [Background] Brokalaki H, Patelarou E, Giakoumidakis K, Kollia Z, Fotos NV, Vivilaki V, Brokalaki E, Chatzistamatiou E, Kallikazaros IE. Translation and validation of the Greek "Minnesota Living with Heart Failure" questionnaire. Hellenic J Cardiol. 2015 Jan-Feb;56(1):10-9. PMID 25701967
- [Background] Evans RA, Singh SJ, Williams JE, Morgan MD. The development of a self-reported version of the chronic heart questionnaire. J Cardiopulm Rehabil Prev. 2011 Nov-Dec;31(6):365-72. doi: 10.1097/HCR.0b013e318228a31a. PMID 21826017